CLINICAL TRIAL: NCT05154578
Title: A Multicentre, Multinational, Parallel Group, Observer-blind, Randomised, Placebo-controlled Study on the Group B Streptococcus Vaccine (GBS-NN/NN2), Investigating the Immunogenicity and Safety of Four Vaccination Regimens in Pregnant Woman, Assessing IgG Specific to AlpN Proteins in Cord Blood and Maternal Blood, and the Safety Profile in Mother and Infant up to 6 Months Post-delivery
Brief Title: Immunogenicity and Safety of GBS-NN/NN2 in Pregnant Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Minervax ApS (Other)
Collaborators: Larix A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: MVX0004
Record Dates: First submitted 2021-11-09; First posted 2021-12-13 (Actual); Results first posted 2025-01-13 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-05

CONDITIONS: Group B Streptococcal Infection
MeSH Terms: conditions — Streptococcal Infections | interventions — Saline Solution

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to one of 5 groups
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Group 1: 4 week dose interval; 2 doses (Experimental): Participants will receive one injection of placebo at 22 (±1) weeks GA, one injection of GBS-NN/NN2 at 26 (±1) weeks GA and one injection of GBS- NN/NN2 at 30 (±1) weeks GA
  Interventions: Biological: GBS-NN/NN2 Vaccine; Biological: Placebo
- Group 2: early intervention; 4 week dose interval; 2 doses (Experimental): Participants will receive one injection of GBS-NN/NN2 at 22 (±1) weeks GA, one injection of GBS-NN/NN2 at 26 (±1) weeks GA and one injection of placebo at 30 (±1) weeks GA
  Interventions: Biological: GBS-NN/NN2 Vaccine; Biological: Placebo
- Group 3: early intervention; 8 week dose interval; 2 doses (Experimental): Participants will receive one injection of GBS-NN/NN2 at 22 (±1) weeks GA, one injection of placebo at 26 (±1) weeks GA and one injection of GBS- NN/NN2 at 30 (±1) weeks GA
  Interventions: Biological: GBS-NN/NN2 Vaccine; Biological: Placebo
- Group 4: single dose (Experimental): Participants will receive one injection of placebo at 22 (±1) weeks GA, one injection of GBS-NN/NN2 at 26 (±1) weeks GA, and one injection of placebo at 30 (±1) weeks GA.
  Interventions: Biological: GBS-NN/NN2 Vaccine; Biological: Placebo
- Group 5: placebo (Placebo Comparator): Participants will receive one injection of placebo at 22, 26 and 30 weeks (±1) GA
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: GBS-NN/NN2 Vaccine — 0.5 mL GBS-NN/NN2 containing 50 μg of GBS-NN and 50 μg of GBS-NN2 and 0.5 mg of aluminium, given by intramuscular injection.
  Arms: Group 1: 4 week dose interval; 2 doses; Group 2: early intervention; 4 week dose interval; 2 doses; Group 3: early intervention; 8 week dose interval; 2 doses; Group 4: single dose
Biological: Placebo — 0.5 mL normal saline given by intramuscular injection
  Other Names: Normal saline

SUMMARY:
This is a phase II, multicentre, multinational, randomized, parallel group, placebo-controlled study of four vaccination regimens in healthy pregnant women. There will be 5 treatment groups; three groups of 60 participants will receive will receive two doses of GBS-NN/NN2 vaccine and one dose of placebo (saline); one group of 60 participants will receive one dose of GBS-NN/NN2 vaccine and two doses of placebo (saline), and one group of 30 participants will receive three doses of placebo (saline).

DETAILED DESCRIPTION:
This is a phase II, multicentre, multinational, randomized, parallel group, placebo-controlled study of four vaccination regimens in healthy pregnant women. There will be 5 treatment groups; Group 1 will receive one injection of placebo at 22 (±1) weeks gestational age (GA), one injection of GBS-NN/NN2 at 26 (±1) weeks GA and one injection of GBS- NN/NN2 at 30 (±1) weeks GA. Group 2 will receive one injection of GBS-NN/NN2 at 22 (±1) weeks GA, one injection of GBS-NN/NN2 at 26 (±1) weeks GA and one injection of placebo at 30 (±1) weeks GA.Group 3 will receive one injection of GBS-NN/NN2 at 22 (±1) weeks GA, one injection of placebo at 26 (±1) weeks GA and one injection of GBS- NN/NN2 at 30 (±1) weeks GA. Group 4 will receive one injection of placebo at 22 (±1) weeks GA, one injection of GBS-NN/NN2 at 26 (±1) weeks GA and one injection of placebo at 30 (±1) weeks GA.

Group 5 will receive an injection of placebo at 22, 26 and 30 weeks (±1) GA. Participants will attend the clinic for assessment visits up to delivery and for a further 3 visits at 28 (±4) days, 90 (±6) days and 180 (±14) days post delivery.

Babies will be also be assessed at delivery, and 28 (±4) days, 90 (±6) days and 180 (±14) days post delivery.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy pregnant woman above the legally defined age of consent at the time of screening
2. Carrying a normal singleton pregnancy, and is at 21+0 to 23+6 weeks GA at the planned tme of the 1st vaccination, as established by first/second trimester ultrasound examination
3. Properly informed about the study and has given written informed consent and parental consent (for her baby) in accordance with the International Conference on Harmonization Good Clinical Practice (ICH GCP) and local legislation prior to the first study intervention
4. Grants access to her own and her baby's study related medical records

Exclusion Criteria

1. Previous vaccination with an investigational Group B Streptococcus (GBS) Vaccine
2. BMI of <17 or >40 at the time of screening
3. Human immunodeficiency virus (HIV), hepatitis B virus (HBV) and/or hepatitis C virus (HCV) positive or positive for syphilis
4. Knowingly carrying, at screening, a malformed or genetically abnormal foetus, incl. renal pelvis dilation, single umbilical artery (screening will be undertaken after the ultrasound conducted for the detection of anomalies)
5. Chronic or pregnancy induced hypertension at screening, >1+ protein in urine regardless of blood pressure or 1+ protein in urine and hypertension
6. Experienced a previous stillbirth prior to going into labour
7. Gestational, type 1 or type 2 diabetes
8. Potential placenta previa as per malformation ultrasound scan
9. Rhesus negative and has anti-D antibodies or other potential harmful antibodies
10. Known or suspected allergies to any components of the vaccine including to aluminium or aminoglycoside antibiotics, or an allergic reaction related to a previous vaccination
11. Fever (temperature >37.9°C) on the day of receiving the first dose or an acute infection in the 7 days before the first dose (the first dose can be delayed if gestational age permits)
12. Received systemic steroids in the 6 weeks before the first dose (inhaled and topical steroids are acceptable)
13. Any lesion (including tattoos) at the planned injection site that will impair the assessment of the injection site
14. Received immunosuppressive medication, chemotherapy or radiotherapy in the 24 weeks before the first dose
15. Received blood, blood products, plasma derivatives or any immunoglobulin preparations in the 12 weeks before the first dose
16. Anaemia, haemoglobin (<10 g/dL, 100 g/L, 6.2 mmol/L)
17. Currently breast feeding
18. Received any investigational medicinal product or vaccine in the 12 weeks or 5 half-lives before the first dose
19. Received an approved vaccine within the 4 weeks before the first dose or expects to receive an approved vaccine during the study. Routine vaccinations recommended during pregnancy (e.g., pertussis and influenza) are permitted but every effort should be made to separate routine vaccinations from the trial vaccinations by at least 7 days.
20. Known or suspected immunodeficiency or cancer (leukaemia, lymphoma), or a family history of congenital or hereditary immunodeficiency
21. History or presence of uncontrolled cardiovascular disease, pulmonary, hepatic, gall bladder or biliary tract, renal, haematological, gastrointestinal, endocrine, immunologic, dermatological, neurological, psychiatric, or autoimmune disease
22. History of, or current drug or alcohol abuse
23. In the opinion of the investigator not suitable for inclusion in the study
24. The pregnancy is considered high risk by treating physicians

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 269 (Actual)
Dates: Start 2022-02-17 (Actual); Primary Completion 2023-04-26 (Actual); Study Completion 2023-10-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeannett Dimsits, Study Director — jdi@minervax.com
Locations (10):
- Denmark (3):
  - Aarhus University Hospital; Skejby, Aarhus
  - Hvidovre University Hospital, Hvidovre
  - Institut for Regional Sundhedsforskning, Kolding
- South Africa (5):
  - ESRU Rahima Moosa Mother and Child Hospital, Johannesburg
  - Shandukani Research Clinic, Johannesburg
  - Wits Vaccines & Infectious Diseases Analytics, Johannesburg
  - Mecru Clinical Research Unit (MeCRU), Pretoria
  - Setshaba Research Centre, Pretoria
- United Kingdom (2):
  - St George's University Hospital, London
  - University Hospital Southampton, Southampton

REFERENCES:
- [Derived] Heath PT, Zuma-Gwala N, Helmig RB, Horne E, Kjaerbye-Thygesen A, Crusell MKW, Nchabeleng M, Strehlau R, Khalil MR, Jones CE, Biccler J, Dimsits J, Johannsson-Lindbom B, Oostvogels L, Madhi SA; MVX0004 study group. Immunogenicity and safety of a group B Streptococcus vaccine (GBS-AlpN) in pregnant women and their infants: a phase 2, multicentre, observer-blind, randomised, placebo-controlled study. Lancet Infect Dis. 2025 Dec 9:S1473-3099(25)00659-0. doi: 10.1016/S1473-3099(25)00659-0. Online ahead of print. PMID 41386262

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first participant first visit took place on 17 February 2022 and the last participant last visit took place on 18 October 2023.
Pre-assignment Details: A total of 269 maternal participants were enrolled in the study and randomised to one of the 5 study groups.
Groups:
- Group 1: 4 Week Dose Interval; 2 Doses: Participants received one injection of placebo at 22 (±1) weeks GA (gestational age), one injection of GBS-NN/NN2 at 26 (±1) weeks GA and one injection of GBS- NN/NN2 at 30 (±1) weeks GA
  GBS-NN/NN2 Vaccine: 0.5 mL GBS-NN/NN2 containing 50 μg of GBS-NN and 50 μg of GBS-NN2 and 0.5 mg of aluminium, given by intramuscular injection.
  Placebo: 0.5 mL normal saline given by intramuscular injection
- Group 2: Early Intervention; 4 Week Dose Interval; 2 Doses: Participants received one injection of GBS-NN/NN2 at 22 (±1) weeks GA, one injection of GBS-NN/NN2 at 26 (±1) weeks GA and one injection of placebo at 30 (±1) weeks GA
  GBS-NN/NN2 Vaccine: 0.5 mL GBS-NN/NN2 containing 50 μg of GBS-NN and 50 μg of GBS-NN2 and 0.5 mg of aluminium, given by intramuscular injection.
  Placebo: 0.5 mL normal saline given by intramuscular injection
- Group 3: Early Intervention; 8 Week Dose Interval; 2 Doses: Participants received one injection of GBS-NN/NN2 at 22 (±1) weeks GA, one injection of placebo at 26 (±1) weeks GA and one injection of GBS- NN/NN2 at 30 (±1) weeks GA
  GBS-NN/NN2 Vaccine: 0.5 mL GBS-NN/NN2 containing 50 μg of GBS-NN and 50 μg of GBS-NN2 and 0.5 mg of aluminium, given by intramuscular injection.
  Placebo: 0.5 mL normal saline given by intramuscular injection
- Group 4: Single Dose: Participants received one injection of placebo at 22 (±1) weeks GA, one injection of GBS-NN/NN2 at 26 (±1) weeks GA, and one injection of placebo at 30 (±1) weeks GA.
  GBS-NN/NN2 Vaccine: 0.5 mL GBS-NN/NN2 containing 50 μg of GBS-NN and 50 μg of GBS-NN2 and 0.5 mg of aluminium, given by intramuscular injection.
  Placebo: 0.5 mL normal saline given by intramuscular injection
- Group 5: Placebo: Participants received one injection of placebo at 22, 26 and 30 weeks (±1) GA
  Placebo: 0.5 mL normal saline given by intramuscular injection
Period: Overall Study
Arm/Group | Group 1: 4 Week Dose Interval; 2 Doses | Group 2: Early Intervention; 4 Week Dose Interval; 2 Doses | Group 3: Early Intervention; 8 Week Dose Interval; 2 Doses | Group 4: Single Dose | Group 5: Placebo
Started | 61 | 59 | 59 | 60 | 30
Number of Live Infant Delivered | 61 | 58 | 58 | 57 | 29
Completed | 59 | 54 | 56 | 52 | 29
Not Completed | 2 | 5 | 3 | 8 | 1
Not completed — Withdrawal by Subject | 2 | 3 | 2 | 4 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 3 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0
Not completed — Relocated to another province | 0 | 0 | 1 | 0 | 1
Not completed — Baby loss | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: 4 Week Dose Interval; 2 Doses | Group 2: Early Intervention; 4 Week Dose Interval; 2 Doses | Group 3: Early Intervention; 8 Week Dose Interval; 2 Doses | Group 4: Single Dose | Group 5: Placebo | Total
Number analyzed (Participants) | 61 | 59 | 59 | 60 | 30 | 269
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 61 | 59 | 59 | 60 | 30 | 269
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.9 (5.26) | 27.5 (4.81) | 27.8 (5.34) | 27.3 (5.37) | 28.3 (6.65) | 27.9 (5.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 59 | 59 | 60 | 30 | 269
  Male | 0 | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 1 | 0 | 1 | 4
  Not Hispanic or Latino | 59 | 59 | 58 | 60 | 29 | 265
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 2 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 44 | 41 | 43 | 44 | 22 | 194
  White | 16 | 18 | 16 | 14 | 8 | 72
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Denmark | 13 | 14 | 12 | 13 | 7 | 59
  United Kingdom | 4 | 3 | 4 | 3 | 1 | 15
  South Africa | 44 | 42 | 43 | 44 | 22 | 195
Height [Mean (Standard Deviation); unit: cm] | 161.7 (7.84) | 162.2 (8.00) | 163.3 (7.58) | 160.5 (6.88) | 160.5 (6.92) | 161.8 (7.53)
Weight [Mean (Standard Deviation); unit: kg] | 71.1 (14.00) | 73.0 (12.11) | 73.6 (14.52) | 70.6 (14.59) | 74.2 (13.38) | 72.3 (13.76)
BMI [Mean (Standard Deviation); unit: kg/m²] | 27.2 (5.28) | 27.9 (5.32) | 27.6 (5.35) | 27.5 (5.57) | 28.8 (5.38) | 27.7 (5.36)

OUTCOME MEASURES:

1. Primary Outcome: Concentrations of Immunoglobulin (Ig) G Antibodies Specific to the AlpN Proteins in μg/mL in Cord Blood From Each Baby
Description: Concentrations of IgG antibodies specific to the AlpN proteins in μg/mL in cord blood from each baby at birth.
Time Frame: Delivery
Population: Baby Immunogenicicty Set : babies with at least one evaluable sample.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Groups:
- Group 1: 4 Week Dose Interval; 2 Doses (Infant Participants): Infants of participants from group 1, who received one injection of placebo at 22 (±1) weeks GA, one injection of GBS-NN/NN2 at 26 (±1) weeks GA and one injection of GBS- NN/NN2 at 30 (±1) weeks GA
- Group 2: Early Intervention; 4 Week Dose Interval; 2 Doses (Infant Participants): Infants of participants from group 2, who received one injection of GBS-NN/NN2 at 22 (±1) weeks GA, one injection of GBS-NN/NN2 at 26 (±1) weeks GA and one injection of placebo at 30 (±1) weeks GA
- Group 3: Early Intervention; 8 Week Dose Interval; 2 Doses (Infant Participants): Infants of participant of group 3, who received one injection of GBS-NN/NN2 at 22 (±1) weeks GA, one injection of placebo at 26 (±1) weeks GA and one injection of GBS- NN/NN2 at 30 (±1) weeks GA
- Group 4: Single Dose (Infant Participants): Infants of participants from group 4, who received one injection of placebo at 22 (±1) weeks GA, one injection of GBS-NN/NN2 at 26 (±1) weeks GA, and one injection of placebo at 30 (±1) weeks GA
- Group 5: Placebo (Infant Participants): Infant of participants from group 5, who received one injection of placebo at 22, 26 and 30 weeks (±1) GA
Arm/Group | Group 1: 4 Week Dose Interval; 2 Doses (Infant Participants) | Group 2: Early Intervention; 4 Week Dose Interval; 2 Doses (Infant Participants) | Group 3: Early Intervention; 8 Week Dose Interval; 2 Doses (Infant Participants) | Group 4: Single Dose (Infant Participants) | Group 5: Placebo (Infant Participants)
Number analyzed (Participants) | 43 | 47 | 47 | 37 | 20
μg/mL
  Alp1N: number analyzed (Participants) | 41 | 45 | 43 | 34 | 20
  Alp1N | 11.12 (236.7) | 5.52 (183.9) | 7.95 (261.6) | 3.51 (565.2) | 0.07 (102.2)
  Alp2N: number analyzed (Participants) | 36 | 43 | 41 | 36 | 20
  Alp2N | 7.93 (164.0) | 5.32 (280.9) | 5.46 (445.7) | 3.39 (717.6) | 0.04 (112.9)
  AlpCN: number analyzed (Participants) | 36 | 47 | 44 | 35 | 20
  AlpCN | 8.85 (246.7) | 6.71 (337.4) | 7.39 (374.6) | 3.10 (682.0) | 0.06 (137.5)
  RibN: number analyzed (Participants) | 38 | 45 | 45 | 36 | 20
  RibN | 3.67 (157.6) | 1.76 (434.2) | 3.23 (283.3) | 1.28 (520.6) | 0.06 (129.4)

2. Secondary Outcome: Injection Site Reactions in the Mother
Description: Number of participants with solicited injection site reactions following vaccination
Time Frame: 7 days following each injection
Measure: Number; unit: participants
Arm/Group | Group 1: 4 Week Dose Interval; 2 Doses | Group 2: Early Intervention; 4 Week Dose Interval; 2 Doses | Group 3: Early Intervention; 8 Week Dose Interval; 2 Doses | Group 4: Single Dose | Group 5: Placebo
Number analyzed (Participants) | 61 | 59 | 59 | 60 | 30
participants
  Redness : 0 - 2.4 cm | 7 | 5 | 9 | 5 | 5
  Redness : 2.5 - 5.0 cm | 2 | 1 | 2 | 0 | 0
  Redness : 5.1 - 10.0 cm | 0 | 1 | 0 | 0 | 0
  Redness : >10 cm | 0 | 0 | 0 | 0 | 0
  Swelling : Palpable "firmness" only | 14 | 10 | 9 | 6 | 1
  Swelling : 0 - 2.4 cm | 5 | 2 | 2 | 2 | 0
  Swelling : 2.5 - 5.0 cm | 0 | 2 | 0 | 0 | 0
  Swelling : 5.1 - 10.0 cm | 0 | 0 | 0 | 0 | 0
  Tenderness: Mild | 14 | 17 | 18 | 16 | 3
  Tenderness: Moderate | 15 | 12 | 13 | 10 | 1
  Tenderness: Severe | 0 | 0 | 1 | 0 | 0
  Itching | 23 | 20 | 15 | 14 | 4
  Pain: Mild | 35 | 35 | 34 | 24 | 3
  Pain: Moderate | 3 | 3 | 2 | 0 | 0
  Pain: Severe | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Adverse Events Following the Vaccinations in the Mother
Description: Number of participants with solicited and other adverse events following the vaccinations
Time Frame: To Day 84
Measure: Number; unit: participants
Arm/Group | Group 1: 4 Week Dose Interval; 2 Doses | Group 2: Early Intervention; 4 Week Dose Interval; 2 Doses | Group 3: Early Intervention; 8 Week Dose Interval; 2 Doses | Group 4: Single Dose | Group 5: Placebo
Number analyzed (Participants) | 61 | 59 | 59 | 60 | 30
participants | 56 | 54 | 57 | 56 | 26

4. Secondary Outcome: Clinically Significant Abnormal Laboratory Tests in the Mother
Description: Number of participants with clinically significant abnormal laboratory tests in the mother
Time Frame: To Day 84
Measure: Number; unit: participants
Arm/Group | Group 1: 4 Week Dose Interval; 2 Doses | Group 2: Early Intervention; 4 Week Dose Interval; 2 Doses | Group 3: Early Intervention; 8 Week Dose Interval; 2 Doses | Group 4: Single Dose | Group 5: Placebo
Number analyzed (Participants) | 61 | 59 | 59 | 60 | 30
participants | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Clinically Significant Changes in Vital Signs in the Mother
Description: Number of participants with clinically significant changes in vital signs (heart rate, blood pressure, oral temperature) in the mother
Time Frame: To Day 84
Measure: Number; unit: participants
Arm/Group | Group 1: 4 Week Dose Interval; 2 Doses | Group 2: Early Intervention; 4 Week Dose Interval; 2 Doses | Group 3: Early Intervention; 8 Week Dose Interval; 2 Doses | Group 4: Single Dose | Group 5: Placebo
Number analyzed (Participants) | 61 | 59 | 59 | 60 | 30
participants | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Clinically Significant Changes in Physical Examination in the Mother
Description: Number of participants with clinically significant changes in physical examination in the mother
Time Frame: To Day 84
Measure: Number; unit: participants
Arm/Group | Group 1: 4 Week Dose Interval; 2 Doses | Group 2: Early Intervention; 4 Week Dose Interval; 2 Doses | Group 3: Early Intervention; 8 Week Dose Interval; 2 Doses | Group 4: Single Dose | Group 5: Placebo
Number analyzed (Participants) | 61 | 59 | 59 | 60 | 30
participants | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: Gestational Age
Description: Gestational age at birth
Time Frame: Delivery
Population: Baby safety analysis set
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Group 1: 4 Week Dose Interval; 2 Doses (Infant Participants) | Group 2: Early Intervention; 4 Week Dose Interval; 2 Doses (Infant Participants) | Group 3: Early Intervention; 8 Week Dose Interval; 2 Doses (Infant Participants) | Group 4: Single Dose (Infant Participants) | Group 5: Placebo (Infant Participants)
Number analyzed (Participants) | 61 | 58 | 58 | 57 | 29
weeks | 38.7 (2.88) | 38.9 (2.39) | 38.9 (2.30) | 38.8 (2.37) | 39.4 (1.45)

8. Secondary Outcome: Weight of the Baby
Description: Weight of the baby
Time Frame: Delivery
Population: Baby safety analysis set
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Group 1: 4 Week Dose Interval; 2 Doses (Infant Participants) | Group 2: Early Intervention; 4 Week Dose Interval; 2 Doses (Infant Participants) | Group 3: Early Intervention; 8 Week Dose Interval; 2 Doses (Infant Participants) | Group 4: Single Dose (Infant Participants) | Group 5: Placebo (Infant Participants)
Number analyzed (Participants) | 61 | 58 | 58 | 57 | 29
grams | 3165.4 (585.45) | 3086.5 (679.50) | 3230.1 (638.71) | 2955.3 (598.35) | 3272.4 (629.20)

9. Secondary Outcome: Length of the Baby
Description: Length of the baby
Time Frame: Delivery
Population: Baby safety analysis set
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Group 1: 4 Week Dose Interval; 2 Doses (Infant Participants) | Group 2: Early Intervention; 4 Week Dose Interval; 2 Doses (Infant Participants) | Group 3: Early Intervention; 8 Week Dose Interval; 2 Doses (Infant Participants) | Group 4: Single Dose (Infant Participants) | Group 5: Placebo (Infant Participants)
Number analyzed (Participants) | 61 | 58 | 58 | 57 | 29
centimeters | 50.3 (3.59) | 49.9 (2.96) | 49.3 (4.88) | 48.9 (4.42) | 49.7 (4.45)

10. Secondary Outcome: Head Circumference of the Baby
Description: Head circumference of the baby
Time Frame: Delivery
Population: Baby safety analysis set
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Group 1: 4 Week Dose Interval; 2 Doses (Infant Participants) | Group 2: Early Intervention; 4 Week Dose Interval; 2 Doses (Infant Participants) | Group 3: Early Intervention; 8 Week Dose Interval; 2 Doses (Infant Participants) | Group 4: Single Dose (Infant Participants) | Group 5: Placebo (Infant Participants)
Number analyzed (Participants) | 61 | 58 | 58 | 57 | 29
centimeters | 34.4 (1.83) | 34.3 (1.68) | 33.8 (2.49) | 34.0 (2.19) | 34.8 (1.60)

11. Secondary Outcome: Apgar Score in the Baby
Description: Apgar score in the baby (Appearance; Pulse; Grimace response; Activity; Respiration).
  Range 0 to 10 where high scores are good and low scores are bad.
Time Frame: 1, 5 and 10 minutes
Population: Baby safety analysis set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group 1: 4 Week Dose Interval; 2 Doses (Infant Participants) | Group 2: Early Intervention; 4 Week Dose Interval; 2 Doses (Infant Participants) | Group 3: Early Intervention; 8 Week Dose Interval; 2 Doses (Infant Participants) | Group 4: Single Dose (Infant Participants) | Group 5: Placebo (Infant Participants)
Number analyzed (Participants) | 61 | 58 | 58 | 57 | 29
score on a scale
  APGAR score at 1 minute | 8.8 (1.39) | 9.0 (0.91) | 8.8 (1.00) | 8.9 (1.38) | 8.8 (1.22)
  APGAR score at 5 minutes | 9.7 (1.34) | 9.8 (0.54) | 9.8 (0.60) | 9.9 (0.32) | 9.8 (0.62)
  APGAR score at 10 minutes | 9.9 (0.29) | 9.9 (0.28) | 9.9 (0.33) | 9.9 (0.29) | 10.0 (0.00)

12. Secondary Outcome: Concentrations of IgG Antibodies Specific to the AlpN Proteins in μg/mL in Maternal Blood
Description: Concentrations of IgG antibodies specific to the AlpN proteins in μg/mL in maternal blood
Time Frame: Delivery
Population: Baby Immunogenicicty Set : babies with at least one evaluable sample.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Group 1: 4 Week Dose Interval; 2 Doses | Group 2: Early Intervention; 4 Week Dose Interval; 2 Doses | Group 3: Early Intervention; 8 Week Dose Interval; 2 Doses | Group 4: Single Dose | Group 5: Placebo
Number analyzed (Participants) | 61 | 59 | 59 | 60 | 30
μg/mL
  Alp1N: number analyzed (Participants) | 56 | 48 | 54 | 52 | 27
  Alp1N | 40.57 (271.0) | 15.81 (295.1) | 32.91 (322.2) | 12.38 (604.4) | 1.03 (85.3)
  Alp2N: number analyzed (Participants) | 56 | 45 | 49 | 47 | 28
  Alp2N | 61.69 (384.9) | 32.74 (275.1) | 39.54 (239.9) | 18.96 (491.4) | 1.02 (95.9)
  AlpCN: number analyzed (Participants) | 58 | 52 | 54 | 51 | 27
  AlpCN | 48.11 (314.7) | 25.17 (328.6) | 27.53 (332.7) | 16.38 (482.6) | 1.10 (86.4)
  RibN: number analyzed (Participants) | 56 | 51 | 52 | 55 | 23
  RibN | 25.55 (323.2) | 10.97 (305.5) | 20.08 (473.4) | 8.68 (614.4) | 0.92 (74.4)

13. Secondary Outcome: Concentrations of IgG Antibodies Specific to the AlpN Proteins in μg/mL in Blood From Each Baby
Description: Concentrations of IgG antibodies specific to the AlpN proteins in μg/mL in blood from each baby
Time Frame: 1 month, 3 months
Population: Baby Immunogenicicty Set : babies with at least one evaluable sample.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Group 1: 4 Week Dose Interval; 2 Doses (Infant Participants) | Group 2: Early Intervention; 4 Week Dose Interval; 2 Doses (Infant Participants) | Group 3: Early Intervention; 8 Week Dose Interval; 2 Doses (Infant Participants) | Group 4: Single Dose (Infant Participants) | Group 5: Placebo (Infant Participants)
Number analyzed (Participants) | 43 | 47 | 47 | 37 | 20
μg/mL
  Alp1N: At 1 month of age: number analyzed (Participants) | 42 | 46 | 41 | 35 | 19
  Alp1N: At 1 month of age | 4.81 (419.4) | 2.92 (184.7) | 7.02 (116.3) | 1.72 (983.6) | 0.05 (424.7)
  Alp1N: At 3 months of age: number analyzed (Participants) | 43 | 43 | 44 | 34 | 20
  Alp1N: At 3 months of age | 1.91 (270.3) | 1.24 (149.0) | 2.26 (152.6) | 0.54 (515.7) | 0.03 (127.2)
  Alp2N: At 1 month of age: number analyzed (Participants) | 40 | 43 | 38 | 33 | 20
  Alp2N: At 1 month of age | 4.25 (379.8) | 2.87 (281.3) | 3.91 (283.4) | 1.43 (916.8) | 0.05 (534.0)
  Alp2N: At 3 months of age: number analyzed (Participants) | 39 | 39 | 40 | 29 | 20
  Alp2N: At 3 months of age | 1.73 (239.6) | 1.05 (256.2) | 1.37 (247.2) | 0.59 (427.3) | 0.02 (102.0)
  AlpCN: At 1 month of age: number analyzed (Participants) | 42 | 45 | 43 | 35 | 20
  AlpCN: At 1 month of age | 4.90 (495.8) | 3.44 (264.8) | 4.64 (399.0) | 1.50 (1065.8) | 0.07 (384.9)
  AlpCN: At 3 months of age: number analyzed (Participants) | 43 | 43 | 44 | 34 | 20
  AlpCN: At 3 months of age | 1.92 (289.2) | 1.15 (323.8) | 1.67 (214.1) | 0.49 (436.0) | 0.03 (106.5)
  RibN: At 1 month of age: number analyzed (Participants) | 42 | 46 | 43 | 35 | 20
  RibN: At 1 month of age | 2.46 (190.5) | 1.13 (223.6) | 2.13 (264.1) | 0.77 (560.9) | 0.05 (237.2)
  RibN: At 3 months of age: number analyzed (Participants) | 43 | 43 | 44 | 34 | 20
  RibN: At 3 months of age | 0.88 (190.2) | 0.45 (219.1) | 0.78 (271.9) | 0.22 (465.2) | 0.03 (92.1)

ADVERSE EVENTS:
Time Frame: Treatment-emergent Adverse Events (TEAEs) in the mother were assessed from the time of informed consent until Day 84. From delivery onwards, only Medically attended adverse events (MAAEs), Adverse events of special interest (AESIs) and Serious adverse events (SAEs) were assessed until the end of study (corresponding to 166-194 days post-delivery). For the infants, all AEs were assessed for the first 28 days of life. Afterward, only MAAEs, AESIs and SAEs were assessed until the end of study.
Description: Solicited local and systemic reactions were collected in electronic diaries up to 7 days following each administered vaccination. In addition, other AEs, i.e., unsolicited AEs, including MAAEs, SAEs, concomitant medication or vaccines were to be recorded in the electronic diary.
  AEs were also collected following laboratory safety tests, physical examinations and vital signs performed at the study visits.
Groups:
- Group 1 (Mothers): 4 Week Dose Interval; 2 Doses: Participants received one injection of placebo at 22 (±1) weeks GA (gestational age), one injection of GBS-NN/NN2 at 26 (±1) weeks GA and one injection of GBS- NN/NN2 at 30 (±1) weeks GA
  GBS-NN/NN2 Vaccine: 0.5 mL GBS-NN/NN2 containing 50 μg of GBS-NN and 50 μg of GBS-NN2 and 0.5 mg of aluminium, given by intramuscular injection.
  Placebo: 0.5 mL normal saline given by intramuscular injection
- Group 2 (Mothers): Early Intervention; 4 Week Dose Interval; 2 Doses: Participants received one injection of GBS-NN/NN2 at 22 (±1) weeks GA, one injection of GBS-NN/NN2 at 26 (±1) weeks GA and one injection of placebo at 30 (±1) weeks GA
  GBS-NN/NN2 Vaccine: 0.5 mL GBS-NN/NN2 containing 50 μg of GBS-NN and 50 μg of GBS-NN2 and 0.5 mg of aluminium, given by intramuscular injection.
  Placebo: 0.5 mL normal saline given by intramuscular injection
- Group 3 (Mothers): Early Intervention; 8 Week Dose Interval; 2 Doses: Participants received one injection of GBS-NN/NN2 at 22 (±1) weeks GA, one injection of placebo at 26 (±1) weeks GA and one injection of GBS- NN/NN2 at 30 (±1) weeks GA
  GBS-NN/NN2 Vaccine: 0.5 mL GBS-NN/NN2 containing 50 μg of GBS-NN and 50 μg of GBS-NN2 and 0.5 mg of aluminium, given by intramuscular injection.
  Placebo: 0.5 mL normal saline given by intramuscular injection
- Group 4 (Mothers): Single Dose: Participants received one injection of placebo at 22 (±1) weeks GA, one injection of GBS-NN/NN2 at 26 (±1) weeks GA, and one injection of placebo at 30 (±1) weeks GA.
  GBS-NN/NN2 Vaccine: 0.5 mL GBS-NN/NN2 containing 50 μg of GBS-NN and 50 μg of GBS-NN2 and 0.5 mg of aluminium, given by intramuscular injection.
  Placebo: 0.5 mL normal saline given by intramuscular injection
- Group 5 (Mothers): Placebo: Participants received one injection of placebo at 22, 26 and 30 weeks (±1) GA
  Placebo: 0.5 mL normal saline given by intramuscular injection
- Group 1 (Infants): 4 Week Dose Interval; 2 Doses: Infants of participants from group 1, who received one injection of placebo at 22 (±1) weeks GA, one injection of GBS-NN/NN2 at 26 (±1) weeks GA and one injection of GBS- NN/NN2 at 30 (±1) weeks GA
- Group 2 (Infants): Early Intervention; 4 Week Dose Interval; 2 Doses: Infants of participants from group 2, who received one injection of GBS-NN/NN2 at 22 (±1) weeks GA, one injection of GBS-NN/NN2 at 26 (±1) weeks GA and one injection of placebo at 30 (±1) weeks GA
- Group 3 (Infants): Early Intervention; 8 Week Dose Interval; 2 Doses: Infants of participant of group 3, who received one injection of GBS-NN/NN2 at 22 (±1) weeks GA, one injection of placebo at 26 (±1) weeks GA and one injection of GBS- NN/NN2 at 30 (±1) weeks GA
- Group 4 (Infants): Single Dose: Infants of participants from group 4, who received one injection of placebo at 22 (±1) weeks GA, one injection of GBS-NN/NN2 at 26 (±1) weeks GA, and one injection of placebo at 30 (±1) weeks GA
- Group 5 (Infants): Placebo: Infant of participants from group 5, who received one injection of placebo at 22, 26 and 30 weeks (±1) GA
Arm/Group | Group 1 (Mothers): 4 Week Dose Interval; 2 Doses | Group 2 (Mothers): Early Intervention; 4 Week Dose Interval; 2 Doses | Group 3 (Mothers): Early Intervention; 8 Week Dose Interval; 2 Doses | Group 4 (Mothers): Single Dose | Group 5 (Mothers): Placebo | Group 1 (Infants): 4 Week Dose Interval; 2 Doses | Group 2 (Infants): Early Intervention; 4 Week Dose Interval; 2 Doses | Group 3 (Infants): Early Intervention; 8 Week Dose Interval; 2 Doses | Group 4 (Infants): Single Dose | Group 5 (Infants): Placebo
All-Cause Mortality (participants affected / at risk) | 0/61 | 0/59 | 0/59 | 0/60 | 0/30 | 2/61 | 2/58 | 1/58 | 3/57 | 1/29
Serious Adverse Events (participants affected / at risk) | 23/61 | 12/59 | 20/59 | 25/60 | 14/30 | 15/61 | 13/58 | 16/58 | 17/57 | 7/29
Other Adverse Events (participants affected / at risk) | 56/61 | 54/59 | 57/59 | 56/60 | 26/30 | 43/61 | 38/58 | 38/58 | 45/57 | 21/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (Mothers): 4 Week Dose Interval; 2 Doses (N=61) | Group 2 (Mothers): Early Intervention; 4 Week Dose Interval; 2 Doses (N=59) | Group 3 (Mothers): Early Intervention; 8 Week Dose Interval; 2 Doses (N=59) | Group 4 (Mothers): Single Dose (N=60) | Group 5 (Mothers): Placebo (N=30) | Group 1 (Infants): 4 Week Dose Interval; 2 Doses (N=61) | Group 2 (Infants): Early Intervention; 4 Week Dose Interval; 2 Doses (N=58) | Group 3 (Infants): Early Intervention; 8 Week Dose Interval; 2 Doses (N=58) | Group 4 (Infants): Single Dose (N=57) | Group 5 (Infants): Placebo (N=29)
Foetal distress syndrome (Pregnancy, puerperium and perinatal conditions) | 8 (8) | 2 (2) | 5 (5) | 12 (12) | 7 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 3 (3) | 2 (2) | 4 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gestational hypertension (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 1 (1) | 4 (4) | 4 (4) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prolonged labour (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 1 (1) | 3 (3) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Premature delivery (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 3 (3) | 2 (2) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foetal death (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 4 (4) | 5 (5) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foetal Growth restriction (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HELLP syndrome (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oligohydramnios (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Postpartum haemorrhage (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
False labour (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foetal hypokinesia (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gestational diabetes (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intrapartum haemorrhage (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Placenta praevia (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Premature labour (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Premature rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abortion threatened (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Amniorrhoea (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cephalo-pelvic disproportion (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Failed induction of labour (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foetal macrosomia (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foetal vascular malperfusion (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large for dates baby (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Premature separation of placenta (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prolonged pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prolonged rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retroplacental haematoma (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uterine hypotonus (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhage in pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meconium in amniotic fluid (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Placental insufficiency (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Amniotic cavity infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacterial vaginosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Endometritis decidual (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Escherichia infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Postpartum sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Beta haemolytic streptococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Postoperative wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection enterococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bradycardia foetal (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Perineal injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney inury (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertensive emergency (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foetal monitoring abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Artificial rupture of membranes (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Jaundice neonatal (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 5 (5) | 3 (3) | 6 (7) | 0 (0)
Low birth weight baby (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 5 (5) | 3 (3) | 2 (2) | 0 (0)
Premature baby (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 3 (3) | 0 (0)
Stillbirth (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 3 (3) | 1 (1)
Sepsis neonatal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 2 (2) | 4 (9) | 1 (1)
Talipes (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Birth mark (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cleft palate (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Congenital skin dimples (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epidermolysis bullosa (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hydrocele (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypospadias (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Patent ductus arteriosus (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Supernumerary nipple (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ventricular septal defect (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infantile fibromatosis (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bone metabolism disorder (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Congenital naevus (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Weight decrease neonatal (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small for dates baby (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Bacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fungal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neonatal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchiolitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Lower respiratory tract infection viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Meningitis neonatal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neonatal pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chronic respiratory disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neonatal respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Neonatal respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (4) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Transient tachypnoea of the newborn (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchopulmonary dysplasia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Meconium aspiration syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper airway obstruction (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Underweight (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Neonatal hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Weight gain poor (Metabolism and nutrition disorders) | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaemia neonatal (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (6) | 0 (0)
Thrombocytopenia neonatal (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Prerenal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Necrotising enterocolitis neonatal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Food protein-induced enterocolitis syndrome (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ileus paralytic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Necrotising colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Body height below normal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Tympanometry abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac murmur (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intraventricular haemorrhage neonatal (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Encephalopathy neonatal (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intraventricular haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Retinopathy of prematurity (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Developmental regression (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Drug withdrawal syndrome neonatal (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (Mothers): 4 Week Dose Interval; 2 Doses (N=61) | Group 2 (Mothers): Early Intervention; 4 Week Dose Interval; 2 Doses (N=59) | Group 3 (Mothers): Early Intervention; 8 Week Dose Interval; 2 Doses (N=59) | Group 4 (Mothers): Single Dose (N=60) | Group 5 (Mothers): Placebo (N=30) | Group 1 (Infants): 4 Week Dose Interval; 2 Doses (N=61) | Group 2 (Infants): Early Intervention; 4 Week Dose Interval; 2 Doses (N=58) | Group 3 (Infants): Early Intervention; 8 Week Dose Interval; 2 Doses (N=58) | Group 4 (Infants): Single Dose (N=57) | Group 5 (Infants): Placebo (N=29)
Urinary tract infection (Infections and infestations) | 15 (17) | 13 (16) | 8 (9) | 14 (16) | 7 (8) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 9 (10) | 5 (5) | 9 (9) | 6 (7) | 5 (6) | 15 (18) | 8 (8) | 11 (12) | 13 (15) | 7 (8)
Gastroenteritis (Infections and infestations) | 1 (1) | 4 (5) | 1 (1) | 2 (3) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Vulvovaginal candidiasis (Infections and infestations) | 3 (3) | 2 (3) | 2 (2) | 6 (6) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Streptococcal urinary tract infection (Infections and infestations) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foetal hypokinesia (Pregnancy, puerperium and perinatal conditions) | 4 (5) | 4 (6) | 7 (7) | 2 (4) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gestational hypertension (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 2 (2) | 4 (4) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prolonged pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uterine contractions during pregnancy (Pregnancy, puerperium and perinatal conditions) | 4 (4) | 1 (1) | 1 (2) | 3 (4) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 4 (5) | 6 (6) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 6 (7) | 2 (2) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 8 (8) | 7 (9) | 5 (5) | 4 (4) | 4 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 3 (3) | 2 (3) | 4 (4) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 2 (2) | 3 (3) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 5 (6) | 5 (5) | 3 (5) | 4 (4) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 4 (4) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 3 (5) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 4 (4) | 3 (3) | 2 (2) | 3 (3) | 1 (4) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 4 (5) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 2 (2)
Hypertension (Vascular disorders) | 2 (2) | 0 (0) | 4 (5) | 1 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Jaundice Neonatal (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 4 (4) | 5 (6) | 3 (3) | 5 (5)
Low birth weight baby (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 4 (4) | 2 (2)
Small for dates baby (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 2 (2) | 4 (4) | 0 (0)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 3 (3) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 2 (2)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 2 (2) | 3 (3) | 2 (2)
COVID-19 (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 2 (2)
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 3 (3) | 3 (3) | 1 (1) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 4 (4) | 2 (2) | 2 (2)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 3 (3) | 2 (2) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-04-14): https://cdn.clinicaltrials.gov/large-docs/78/NCT05154578/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-30): https://cdn.clinicaltrials.gov/large-docs/78/NCT05154578/SAP_001.pdf